CLINICAL TRIAL: NCT05902208
Title: Contribution of an Antiviral Drug (Valaciclovir) in the Treatment of Generalized Periodontitis (Stage III or IV and Grade A, B or C): Prospective, Randomized and Double Blind Clinical Trial
Acronym: HERPARO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-API-02
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Periodontitis Chronic Generalized Severe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valaciclovir (Experimental)
  Interventions: Drug: Antiviral treatment with conventional non-surgical treatment
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo with conventional non-surgical treatment

INTERVENTIONS:
Drug: Antiviral treatment with conventional non-surgical treatment — Valaciclovir, a antiviral treatment will be added to the conventional non-surgical treatment of generalized periodontitis. One gram per day will be administered during 28 days.
  Arms: Valaciclovir
Drug: Placebo with conventional non-surgical treatment — Placebo of valaciclovir (same composition, without active substance) will be added to the conventional non-surgical treatment of generalized periodontitis. One gram a day will be administered during 28 days.
  Arms: Placebo

SUMMARY:
Periodontitis is an inflammatory pathology that destroys periodontitis and causes tooth loosening. Its high incidence, combined with very high oral and systemic morbidity, places this pathology at the heart of global public health priorities. The current therapeutic management of periodontitis is not satisfactory because it often leads to a stabilization of the disease, marked by frequent recurrences, especially severe forms. Improving the treatment of patients with periodontitis is therefore an essential priority.

If gingival bacterial dysbiosis is a major contributing factor, this model has clinical-biological limitations that suggest that other etiological factors are involved, and worsen the pathology. In particular, the literature provides clear evidence that periodontal lesions are mostly infected with Herpes EBV, CMV and HSV-1 viruses and that periodontal infection with these viruses is very directly correlated with disease progression (severity). In addition, our work provides new cellular and molecular data that demonstrate mechanisms of active EBV infection of cells and periodontal structures, and highlight inflammatory and necrotic effects associated with this infection. Given these observations and the high pathogenicity of herpes viruses, all known to be powerful inflammatory, lytic and immunomodulatory agents, it seems difficult not to evoke a direct etiopathogenic role of these viruses capable of acting synergistically with periodontopathogenic bacteria.

In this context, the use of an antiviral appears as a very attractive therapeutic proposal to effectively treat periodontitis in combination with conventional treatments. This original and innovative proposal can also be easily and quickly validated in a randomized therapeutic trial through the availability of antiviral molecules that are non-toxic and very specific to human herpes viruses that are derivatives of aciclovir.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18
* Diagnosis of periodontitis induced by bacterial biofilms of dental plaque, generalized, stage III or IV and grade A, B or C
* Patients of childbearing age will need to use an effective method of contraception for the duration of their study participation
* Signature of informed consent
* Membership of a social security scheme

Exclusion criteria:

* Necrotizing periodontitis
* Pathologies requiring prophylactic antibiotics therapy (which may influence treatment)
* Non-surgical periodontal treatment completed within 6 months prior to inclusion
* Patients with enhanced protection, namely lactating women, persons deprived of liberty by judicial or administrative decision, person over 18 under legal protection
* Patients who do not accept conventional therapy (gingival debridement not covered by the social security system (performed in each center)
* Periodontitis as a direct manifestation of systemic diseases
* Major systemic pathologies (diabetes, HIV, cancers, immunocompromised patients)
* Negative serology for EBV: a blood test will be performed. the results will be communicated to the patient by the dental surgeon
* Pregnant woman: a blood pregnancy test will be carried out for women of childbearing age who do not have contraception. Results will be communicated to the patient by the dental surgeon
* Renal failure (creatinine clearance < 60 mL/min)
* Systemic antibiotic therapy or any medication affecting the periodontal environment (systemic antibiotics, antiepileptics, immunosuppressants, calcium inhibitors) taken within 6 months of inclusion
* Nephrotoxic medications (aminoglycosides, organoplatinums, iodized contrast agents, methotrexate, pentamidine, foscarnet, cyclosporine and tacrolimus)
* Hypersensitivity to valaciclovir, aciclovir or one of the excipients
* History of DRESS syndrome under valaciclovir treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Compare the efficacy of antiviral treatment (valaciclovir) with conventional non-surgical treatment (scaling and root planing) to conventional treatment with a placebo for generalized periodontitis (stage III or IV and grade A, B or C) | 28 days after the end of antiviral treatment and 2 months after root surfacing
  Efficacy will be assessed by measuring the periodontal pocket depth using a graduated (in millimeter) and coloured probe used at low pressure (<0.2N) 28 days after the end of antiviral treatment (visit 2) and 2 months after scaling and root planing (visit 3), during the periodontal reassessment visit

SECONDARY OUTCOMES:
Compare the efficacy of valaciclovir associated with conventional treatment to conventional treatment with placebo in the management of generalized periodontitis using a conventional periodontal clinical index, the Bleeding on Probing (BOP). | 6 and 8 months after scaling and root planing
  The Bleeding on Probing (BOP) assesses the gingival inflammation based on gum bleeding after periodontal probing. It corresponds to the number of sites with bleeding divided by the total number of measured sites, expressed as a percentage. This index will be collected from the same tooth that was determined for the primary objective.
Compare the efficacy of valaciclovir associated with conventional treatment to conventional treatment with placebo in the management of generalized periodontitis using a conventional periodontal clinical index, the O'Leary's plaque index (PI). | 6 and 8 months after scaling and root planing
  O'Leary's Plaque Index (PI) measures the amount of plaque on the tooth (hygiene index). It is calculated by dividing the number of sites with plaque by the total number of measured sites, expressed as a percentage. This index will be collected from the same tooth that was determined for the primary objective.
Compare the efficacy of valaciclovir associated with conventional treatment to conventional treatment with placebo in the management of generalized periodontitis using a conventional periodontal clinical index, the Clinical Attachment Level (CAL). | 6 and 8 months after root planing
  The Clinical Attachment Level (CAL) assesses the degree of impairment, by measuring the distance between the bottom of the pocket and the amelo-cemental junction of the tooth, expressed in millimeters. This index will be collected from the same tooth that was determined for the primary objective.
Compare the efficacy of valaciclovir associated with conventional treatment to conventional treatment with placebo in the management of generalized periodontitis using a conventional periodontal clinical index, the periodontal pocket depth after probing | 6 and 8 months after root planing
  The periodontal pocket depth will be measured using a graduated (in millimeter) and coloured probe used at low pressure (<0.2N). This index will be collected from the same tooth that was determined for the primary objective.
Compare changes in the Epstein-Barr Virus (EBV) levels, between the two groups of patients | From the start of treatment (V0) to the end of the follow-up (V5, 8 months)
  The Epstein-Barr Virus (EBV) levels in periodontal sample is measured through quantitative Polymerase Chain Reaction (PCR) of their viral genomes, throughout patient follow-up.
Compare changes in the CytoMegaloVirus (CMV) levels between the two groups of patients | From the start of treatment (V0) to the end of the follow-up (V5, 8 months)
  The CytoMegaloVirus (CMV) levels in periodontal sample is measured through quantitative Polymerase Chain Reaction (PCR) of their viral genomes, throughout patient follow-up.
Compare changes in the Herpes Simplex Virus-1 (HSV-1) levels between the 2 patient groups. | From the start of treatment (V0) to the end of the follow-up (V5, 8 months)
  The Herpes Simplex Virus-1 (HSV-1) levels in periodontal sample is measured through quantitative Polymerase Chain Reaction (PCR) of their viral genomes, throughout patient follow-up.
Compare changes in main bacterial species quantity of the periodontal biofilm (bacterial mapping) between both groups. | Before (V0), at the end (V2) and after the antiviral treatment (V5)
  The twenty bacterial species levels in periodontal sample is measured through quantitative Polymerase Chain Reaction (PCR) of the bacterial genomes, before, at the end and after the antiviral treatment (V0, V2 and V5)
Compare frequency of periodontal surgery from visit (V3) (at periodontal reassessment) between both groups | 2 months after the start of the antiviral treatment (V3)
  Surgery is available from visit 3 (during periodontal reassessment) and is indicated for patients with a good degree of hygiene (PI ≤ 20%) but with persistent pockets (PPS > 5mm) and bleeding at probing
Compare changes of oral health impact on the quality of life of patients between both groups | Before (V0), 2 months (V3) and 8 months (V5) after the start of the antiviral treatment
  The oral health impact on quality of life is based on the Oral Health Impact Profile 14 (OHIP-14) questionnaire, which measures the impact of oral conditions on the well-being and quality of life of the patients. It will be measured before, 2 months and 8 months after the start of the antiviral treatment.
Evaluate the medico-economic impact of valaciclovir used with conventional treatment compared to conventional treatment alone. | From the start of treatment (V0) to the end of the follow-up (V5, 8 months)
  The medico-economic impact is evaluated by the incremental cost-effectiveness ratio by divided the difference in the cost of each strategy to the difference in efficiency (number of patients who had therapeutical surgery during the follow-up period)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Nice, Nice, Alpes Maritimes
  - APHM, Marseille, Bouches Du Rhone
  - CHU de Rennes, Rennes, Ille-et-Vilaine

IPD SHARING:
Plan to Share IPD: No